CLINICAL TRIAL: NCT00436449
Title: A Double Blind, Within Subject, Placebo Controlled Randomised Trial to Investigate the Scar Improvement Efficacy of a Single Intradermal Application of RN1001 (Avotermin) in Female Subjects Undergoing Bilateral Breast Augmentation
Brief Title: RN1001(Avotermin) in Scar Improvement Following Breast Augmentation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RN1001-319-1010
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Mammaplasty; Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avotermin

SUMMARY:
This will be a multi-centre, double-blind, within-subject, placebo controlled randomised trial in female subjects. All subjects will undergo bilateral breast augmentation surgery. Immediately following surgery, each subject will receive 100µl containing 50ng or 200ng of RN1001 per linear centimetre intradermally into both margins of one breast wound, and 100µl of placebo solution per linear centimetre intradermally into both margins of their other breast wound. The allocation of treatment to wound (left or right) will be randomised and double blind.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between 18 and 60 years of age undergoing bilateral breast augmentation through an infra-mammary fold incision who have given written informed consent.
* Weight between 50 and 150kg and a body mass index within the permitted range for their height using Quetelet's index-weight (kg)/height²(m). The permitted index is between 15-55.
* Subjects of child bearing potential who are using method(s) of contraception acceptable to the Investigator and agree to do so from at least the screening visit until 1 month post surgery.
* Subjects where the same implant position will be used for each breast; the implants can be placed in sub-mammary or sub-pectoral pockets.
* Subjects where the same type and size of implant is to be used for each breast.
* Subjects with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol . All laboratory tests must be performed within 28 days prior to Day 0.

Exclusion Criteria:

* Subjects with significant breast asymmetry where this may produce a different length or site of wound, or where there will be a different post-operative tension on the wound.
* Subjects who on direct questioning and physical examination have a history or evidence of hypertrophic or keloid scarring.
* Subjects who have had surgery in the area to be incised within one year of Day 0.
* Subjects with a personal history of a bleeding disorder.
* Subjects with any history of breast malignancy.
* Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Subjects who on direct questioning and/or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing.
* Subjects with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Subjects who are taking, or have taken, any investigational drugs including RN1001 within 3 months prior to the screening visit.
* Subjects who are taking regular, continuous, oral corticosteroid therapy.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects who are or who become pregnant up to and including Day 0 or who are lactating.
* Subjects with diseases or conditions that could in the opinion of the Investigator interfere with the assessment of safety, tolerability and efficacy.
* In the opinion of the Investigator, a subject who is not likely to complete the trial for what ever reason.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2004-12; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Investigator scar assessment
Patient scar assessment
Independent scar assessment

SECONDARY OUTCOMES:
Local tolerance
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Whitby, Principal Investigator — BUPA Hospital Manchester
Locations (7):
- United Kingdom (7):
  - The Fitzwilliam Clinic, Belfast
  - The Grosvenor Nuffield Hospital, Chester
  - Classic Hull & East Riding, Hull
  - Hull Nuffield Hospital, Hull
  - Renovo CTU, Manchester
  - BUPA Hospital, Manchester
  - BUPA North Cheshire Hospital, Warrington